CLINICAL TRIAL: NCT04693962
Title: Fibroblast Growth Factor-23 as a Marker of Acute Kidney Injury After Partial Nephrectomy
Brief Title: FGF23 as a Marker of Acute Kidney Injury
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Nicolas Valls Jimenez, MD, MSc, University of Chile
Other Study IDs: OAIC 868/17
Record Dates: First submitted 2020-12-30; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Acute Kidney Injury; Kidney Ischemia
Keywords: Acute kidney injury; Creatinine; Fibroblast Growth Factor-23
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Partial Nephrectomy (PN): Patients that will undergo PN with a transient and controlled renal ischemia injury using a renal artery clamping.
  Interventions: Diagnostic Test: Plasmatic Fibroblast Growth Factor-23 by means of ELISA
- Hemicolectomy (HC): Patients who will undergo HC, as non-renal ischemia surgery controls, with similar demographic characteristics, but submitted to HC.
  Interventions: Diagnostic Test: Plasmatic Fibroblast Growth Factor-23 by means of ELISA
- Nephrolithotomy (NL): Patients who undergo NL as non-renal ischemia surgery controls but with kidney physical injury
  Interventions: Diagnostic Test: Plasmatic Fibroblast Growth Factor-23 by means of ELISA

INTERVENTIONS:
Diagnostic Test: Plasmatic Fibroblast Growth Factor-23 by means of ELISA — Plasma levels of FGF-23 will be measured by ELISA

SUMMARY:
A partial nephrectomy (PN) preserves renal parenchyma with a proper oncology outcome. PN is performed during transitory ischemia to avoid massive bleeding during tumor resection. Nevertheless, the transitory ischemia might cause an acute kidney injury(AKI). AKI diagnose is based on the increase in plasma creatinine concentration and a decrease in urine output. However, both plasma creatinine concentration and diuresis are useful for the diagnose, but not in the detection of the risk patients. Therefore, there is considerable interest to find a biomarkers of kidney injury that allow clinicians to predict the development of AKI. Hence, we propose Fibroblastic Growth Factor-23 (FGF23) as a novel early biomarker to detect patients in risk to develop postoperative AKI after a PN.

We will conduct an observational and prospective study in three different groups of patients: PN gropup, patients who underwent PN with a transient and controlled renal ischemia injury using a renal artery clamping; Hemicolectomy (HC) group, patients as non-renal ischemia surgery controls, with similar demographic characteristics, but submitted to HC; and Nephrolithotomy (NL) group, patients who underwent NL, as a control of kidney surgery with physical injury.

In each patient, a time curve of plasmatic creatinine, blood urea nitrogen (BUN), and FGF23 were measure.

Our study aims to describe the role of FGF23 as an early biomarker of AKI after PN, where patients are exposed to a controlled ischemic injury.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology physical status (ASA) I or II.
* Normal preoperative plasma creatinine level
* Baseline estimated glomerular filtration rate (eGFR) > 60 ml/min per 1.73 m2.

Exclusion Criteria:

* History of chronic kidney disease
* Anemia
* Alterations in the parathormone or vitamin D axis
* Pregnant women
* Subjects with concomitant use of nephrotoxic drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients with a diagnose that requires any of three surgerys: Partial Nephrectomy, Hemicolectomy, Nephrolithotomy
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Acute Kidney Injury | 72 hours
  Patients that develop postoperative acute kidney injury

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic Universidad de Chile, Santiago, Chile

IPD SHARING:
Plan to Share IPD: No